CLINICAL TRIAL: NCT06782828
Title: Accuracy of FNAC in Diagnosis of Thyroid Nodules
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Abed Abdulmoneim Mohammed, Principal Investigator, Assiut University
Other Study IDs: FNAC in thyroid nodules
Record Dates: First submitted 2023-12-25; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-12

CONDITIONS: Thyroid Nodule
MeSH Terms: conditions — Thyroid Nodule

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: observe results of FNAC — observe results of FNAC and compare it with results of histopathological examination to detect accuracy of FNAC in diagnosis of thyroid nodules.

SUMMARY:
Detection of degree of accuracy of FNAC in diagnosis of thyroid nodules

DETAILED DESCRIPTION:
Accuracy in diagnosis in any case is required, and this is beneficial to the patient and the physician, and with the development that currently exists and the trend to use less invasive techniques, accuracy of FNAC should be studied well.1.Thyroid nodules are common and the principal method of diagnosis is fine-needle aspiration cytology (FNAC).2. Can investigators depend on FNAC alone in diagnosis of thyroid nodule in the future?!3. In this study, investigators will compare the results of (FNAC) versus (Biopsy) in diagnosis of thyroid nodule in AUH , to detect the degree of accuracy of FNAC.4. FNAC is a simple, safe, cost-effective and accurate diagnostic tool for the initial screening of patients with thyroid nodules.5. Background Routine application of fine needle aspiration cytology (FNAC) has decreased unnecessary referral of thyroid nodules for surgical treatment and has also increased the cancer rates found in surgery materials. Success of thyroid FNAC depends on skilled aspiration, skilled cytological interpretation and rational analysis of cytological and clinical data. The aim of this study was to determine the diagnostic accuracy rates of thyroid FNAC results obtained in our hospital.6. The FNAC is a sensitive, specific, and accurate initial diagnostic test for the preoperative evaluation of patients with thyroid swellings in our setting as well. The correlation of cytological and histopathological diagnoses is an important quality assurance method, as it allows cytopathologists to calculate their false-positive and false negative results.7

ELIGIBILITY:
Inclusion Criteria:

1. thyroid disease
2. multinodular
3. single nodule
4. TIRAD 3 or more by US
5. thyroid disease underwent FNAC then surgery
6. all age groups
7. patient fit for surgery

Exclusion Criteria:

1. patients with comorbidities.
2. patients unfit for surgery
3. patients who refused surgery.
4. Patient with no diagnostic FNAC.

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients presented to General Surgery Department with either solitary or multiple suspicious thyroid nodules during time of research.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of true positive results of FNAC after thyroidectomy | 12 days
  Accuracy of FNAC in thyroid nodules compared to surgical specimen histopathological examination
Percentage of malignant thyroid nodules not observed by FNAC | 12 days
  Percentage of malignant thyroid nodules that FNAC fails to detect
Incidence of false negative results by FNAC | 12 days
  False negative that diagnosed by FNAC not malignant but proved malignancy after surgical excision
Percentage of total number of true results of FNAC to the total number of cases | 12 days
  Accuracy of FNAC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Poller DN, Stelow EB, Yiangou C. Thyroid FNAC cytology: can we do it better? Cytopathology. 2008 Feb;19(1):4-10. doi: 10.1111/j.1365-2303.2007.00492.x. Epub 2007 Oct 3. PMID 17916090
- [Background] Bhise SV, Shaikh A, Hippargekar PM, Kothule S. A Prospective Study of Ultrasonographic and FNAC Correlation of Thyroid Swellings with Histopathology. Indian J Otolaryngol Head Neck Surg. 2022 Oct;74(Suppl 2):1942-1948. doi: 10.1007/s12070-020-01922-w. Epub 2020 Jun 24. PMID 36452634
- [Background] Momin MA, Bhuiyan FU, Chakraborty S, Kar NK. FNAC and Its Utility in Solitary Thyroid Nodule and Its Correlation with Histopathological Examination. Mymensingh Med J. 2019 Apr;28(2):356-363. PMID 31086151